CLINICAL TRIAL: NCT05366036
Title: Post Marketing Surveillance Study for Tecfidera (Dimethyl Fumarate) Capsules in Korean Patients With Relapsing-Remitting Multiple Sclerosis
Brief Title: A Study for Tecfidera (Dimethyl Fumarate) Capsules in Korean Participants With Relapsing-Remitting Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: MS0008
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis, Relapsing-remitting
Keywords: MS0008; Dimethyl Fumarate; Multiple sclerosis; Tecfidera; Korean participants
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with MS: Participants with relapsing-remitting MS who are newly prescribed and will start treatment with Tecfidera in a real-world clinical practice setting will be observed prospectively for up to 24 months.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The primary purpose of this study is to evaluate the overall safety and efficacy of Tecfidera (Dimethyl Fumarate) as an oral treatment for Korean participants with relapsing-remitting multiple sclerosis (MS) under routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. The decision by the treating physician to prescribe Tecfidera is made before participating in the post marketing surveillance (PMS)
2. A participant data release consent form is signed and dated by the participant and/or legal representative
3. A Korean participant is diagnosed as relapsing-remitting MS per approved Korean label

Exclusion Criteria:

1. Participants with hypersensitivity to active ingredient or any of the excipients of Tecfidera according to the approved Korean label
2. Participants with unresolved serious infection
3. Participants who are participating in another study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Korean participants with relapsing-remitting MS will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 24 months
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not related to the study drug.
Number of Participants With Adverse Drug Reactions (ADRs) | Up to 24 months
  An ADR is defined as all the adverse and unintended responses which are generated from the normal administration/use of study drugs which are cases of not excluding the casual relationship with the study drug, and which shall be regarded as ADRs in the case the relationship with study drug is not known among AEs reported voluntarily.
Number of Participants With Serious Adverse Events (SAEs) | Up to 24 months
  A SAE is defined as any untoward medical occurrence at any dose that meets any of the following criteria: is fatal or life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; or includes other important medical events.
Number of Participants With Serious Adverse Drug Reactions (SADRs) | Up to 24 months
  SADRs are defined as SAEs considered related to Tecfidera by the treating physician.
Number of Participants With Unexpected AEs | Up to 24 months
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not related to the study drug. Expectedness of events are determined according to the approved local label. Unexpected AE is except for any expectedness of events. An unexpected AE is defined as an AE with a difference in nature, severity, specificity, or outcome, compared to the product licensure/safety notification of the drug.
Number of Participants With Unexpected ADRs | Up to 24 months
  An ADR is defined as all the adverse and unintended responses which are generated from the normal administration/use of study drugs which are cases of not excluding the casual relationship with the study drug, and which shall be regarded as ADRs in the case the relationship with study drug is not known among AEs reported voluntarily. Expectedness of events will be determined according to the approved local label. Unexpected ADR means except for any expected ADR in local label. An unexpected ADR is defined as an ADR with difference in the nature or severity, specificity, or the outcome, compared to the product licensure/notification of the drug.

SECONDARY OUTCOMES:
Annualized Relapse Rate | Up to 24 months
  Annualized relapse rate will be calculated as the total number of relapses experienced divided by the total number of participant-years on study treatment. A relapse is defined as the appearance of a new neurological abnormality, or worsening of previously stable, or improving pre-existing neurological abnormality, separated by at least 30 days from the onset of a preceding clinical demyelinating event.
Percentage of Relapsing Participants | Up to 24 months
  Percentage of relapsing participants will be assessed at the time of 24 months from the first administration of Tecfidera. A relapse is defined as the appearance of a new neurological abnormality, or worsening of previously stable, or improving pre-existing neurological abnormality, separated by at least 30 days from the onset of a preceding clinical demyelinating event.
Number of Gadolinium (Gd) Enhancing Lesions | Up to 24 months
  Number of Gd enhancing lesions will be observed using magnetic resonance imaging (MRI) scans.
Change from Baseline in Participant's Global Efficacy Assessment by the Treating Physician | Up to 24 months
  Global efficacy assessment will be evaluated according to the treating physician's clinical discretion with 3-point rating scale at the time of 24 months from the first administration considering participant's overall condition compared to baseline. The score ranges from 1-3. The 3-point rating scale is classified as: 1=Improvement (symptoms are improved, or it is considered as maintaining effect after administration of Tecfidera). Maintaining effect is defined as it is highly expected that Tecfidera discontinuation worsens symptoms, or the same effect is persistent when the previous drug is replaced by Tecfidera; 2=No change (no changes were seen compared to before administration of Tecfidera without any change in concomitant medication or treatment related to MS; not considered as maintaining effect); 3=Worsening (symptoms are worsened compared to before administration of Tecfidera).

CONTACTS AND LOCATIONS:
Locations (20):
- South Korea (20):
  - Site #20, Cheonan, Chungcheongnam-do
  - Site #15, Ansan, Gyeonggi-do
  - Site #08, Bucheon-si, Gyeonggi-do
  - Site #09, Goyang-si, Gyeonggi-do
  - Site #14, Goyang-si, Gyeonggi-do
  - Site #23, Changwon, Gyeongsangnam-do
  - Site #13, Jinju, Gyeongsangnam-do
  - Site #02, Busan
  - Site #16, Busan
  - Site #01, Daegu
  - Site #17, Daegu
  - Site #07, Daejeon
  - Site #03, Kwangju
  - Site #04, Seoul
  - Site #06, Seoul
  - Site #11, Seoul
  - Site #12, Seoul
  - Site #18, Seoul
  - Site #19, Seoul
  - Site #21, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.